CLINICAL TRIAL: NCT00304070
Title: Treatment of Adrenocortical Tumors With Surgery Plus Lymph Node Dissection and Multiagent Chemotherapy: A Groupwide Phase III Study
Brief Title: Cisplatin-Based Chemotherapy and/or Surgery in Treating Young Patients With Adrenocortical Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAR0332; NCI-2009-00413 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARAR0332; ARAR0332; CDR0000467191; ARAR0332 (Other: Children's Oncology Group); ARAR0332 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stage I Adrenal Cortical Carcinoma AJCC v7; Stage II Adrenal Cortical Carcinoma AJCC v7; Stage III Adrenal Cortical Carcinoma AJCC v7; Stage IV Adrenal Cortical Carcinoma AJCC v7
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Mitotane; Dichlorodiphenyldichloroethane; Ethane; pegfilgrastim

ARMS (3):
- Stratum I (surgery, observation) (Experimental): Patients undergo primary tumor resection and retroperitoneal lymph node sampling followed by observation. Patients who have undergone prior surgery without nodal sampling undergo observation only.
  Interventions: Procedure: Conventional Surgery
- Stratum II (exploratory surgery, observation) (Experimental): Patients undergo primary tumor resection and extended regional lymph node dissection followed by observation. Patients who have undergone prior surgery with simple resection of the primary tumor undergo exploratory surgery with extended regional lymph node dissection followed by observation.
  Interventions: Procedure: Conventional Surgery
- Stratum III (chemotherapy, surgery) (Experimental): Patients receive combination chemotherapy with filgrastim (G-CSF) for up to 30 weeks (10 courses) followed by mitotane alone for an additional 2 months. Some patients undergo surgery after chemotherapy course 2 or 4. Some patients undergo additional surgery after finishing all chemotherapy.
  Interventions: Drug: Cisplatin; Procedure: Conventional Surgery; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Biological: Filgrastim; Drug: Mitotane; Biological: Pegfilgrastim

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Stratum III (chemotherapy, surgery)
Procedure: Conventional Surgery — Patients undergo surgery
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Stratum III (chemotherapy, surgery)
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
  Arms: Stratum III (chemotherapy, surgery)
Biological: Filgrastim — Given subcutaneously
  Other Names: Filgrastim-aafi; Filgrastim-ayow; G-CSF; Neupogen; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tevagrastim
  Arms: Stratum III (chemotherapy, surgery)
Drug: Mitotane — Given orally
  Other Names: (o,p)-DDD; 1, 1-Dichloro-2-(o-chlorophenyl)-2-(p-chlorophenyl)ethane; 1-Chloro-2-[2,2-dichloro-1-(4-chlorophenyl)ethyl]benzene; 2, 2-Bis(2-chlorophenyl-4-chlorophenyl)-1,1-dichloroethane; 2, 4'-Dichlorodiphenyldichloroethane; CB 313; CB-313; Chloditan; Chlodithane; DDD; Ethane, 2-(o-chlorophenyl)-2-(p-chlorophenyl)-1,1-dichloro-; Khloditan; Lisodren; Lysodren; Mytotan; o,p' - DDD; o,p'-DDD; Ortho,para-DDD; WR-13045
  Arms: Stratum III (chemotherapy, surgery)
Biological: Pegfilgrastim — Given subcutaneously
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo
  Arms: Stratum III (chemotherapy, surgery)

SUMMARY:
This phase III clinical trial is studying how well cisplatin-based chemotherapy and/or surgery works in treating young patients with stage I, stage II, stage III or stage IV adrenocortical cancer. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe the outcome of patients with stage I adrenocortical tumor (ACT) treated with surgery alone.

II. Describe the outcome of patients with stage II ACT treated with radical adrenalectomy plus regional retroperitoneal lymph node dissection.

III. Describe the outcome of patients with unresectable or metastatic ACT treated with mitotane and a cisplatin-based chemotherapy regimen.

SECONDARY OBJECTIVES:

I. Determine the feasibility and complications associated with the use of radical adrenalectomy and regional node dissection (RLND) in these patients.

II. Determine the toxicity of mitotane when administered with cisplatin, etoposide, and doxorubicin hydrochloride in patients with residual disease after surgery, inoperable tumors, or metastatic disease at diagnosis.

III. Determine, prospectively, the frequency of tumor spillage during surgery in these patients.

IV. Determine the frequency of lymph node involvement in these patients. V. Compare the incidence and type of germline p53 mutation in non-Brazilian children and children from Southern Brazil.

VI. Characterize the cooperating molecular alterations associated with ACT. VII. Determine the presence of embryonal markers in children with ACT.

OUTLINE:

STRATUM I (stage I disease): Patients undergo primary tumor resection and retroperitoneal lymph node sampling followed by observation. Patients who have undergone prior surgery without nodal sampling undergo observation only.

STRATUM II (stage II disease): Patients undergo primary tumor resection and extended regional lymph node dissection followed by observation. Patients who have undergone prior surgery with simple resection of the primary tumor undergo exploratory surgery with extended regional lymph node dissection followed by observation.

STRATUM III (stage III or IV disease):

INDUCTION CHEMOTHERAPY: Patients receive cisplatin-based chemotherapy comprising oral mitotane four times daily on days 1-21; cisplatin IV over 6 hours on days 1-2; etoposide IV over 1 hour on days 1-3; and doxorubicin hydrochloride IV over 1 hour on days 4-5. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 6 and continuing until blood counts recover OR pegfilgrastim SC once on day 6. Treatment repeats every 21 days for 2-4 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or partial response proceed to surgery. Patients with a complete response proceed directly to continuation chemotherapy.

SURGERY: Patients with stage III disease undergo extended surgery and regional lymph node dissection. Patients with stage IV disease undergo primary tumor resection (if feasible) with regional lymph node dissection and resection of the metastases. Patients then proceed to continuation chemotherapy.

CONTINUATION CHEMOTHERAPY: Patients receive additional cisplatin-based chemotherapy (as in induction chemotherapy) for 4-6 courses followed by mitotane alone for an additional 2 months. Patients with stage IV disease then proceed to additional surgery when feasible.

ADDITIONAL SURGERY: Patients with stage IV disease may undergo additional primary tumor resection with regional lymph node dissection and resection (or re-resection) of the metastases.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adrenocortical carcinoma

  * Newly diagnosed disease within the past 3 weeks
  * Any disease stage allowed
* Lansky performance status 60-100% (for patients ≤ 16 years old)
* Karnofsky performance status 60-100% (for patients > 16 years old)
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age as follows:

  * 0.4 mg/dL (1 month to < 6 months)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to < 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (≥ 16 years of age)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT < 2.5 times ULN
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No previous chemotherapy for adrenocortical carcinoma

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2007-05-03 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, Principal Investigator — Children's Oncology Group
Locations (91):
- United States (81):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Albany Medical Center, Albany, New York
  - University of Rochester, Rochester, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Brazil (2):
  - Boldrini Children's Cancer Center, Campinas, São Paulo
  - Instituto De Oncologia Pediatrica, São Paulo
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Derived] Pinto EM, Maxwell KN, Halalsheh H, Phillips A, Powers J, MacFarland S, Walsh MF, Breen K, Formiga MN, Kriwacki R, Nichols KE, Mostafavi R, Wang J, Clay MR, Rodriguez-Galindo C, Ribeiro RC, Zambetti GP. Clinical and Functional Significance of TP53 Exon 4-Intron 4 Splice Junction Variants. Mol Cancer Res. 2022 Feb;20(2):207-216. doi: 10.1158/1541-7786.MCR-21-0583. Epub 2021 Oct 21. PMID 34675114
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1: Stage I Disease (surgery, observation)
- Stratum 2: Stage II Disease (surgery, observation)
- Stratum 3: Stage III OR IV Disease (chemotherapy)
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Started | 24 | 15 | 39
Completed | 21 | 8 | 27
Not Completed | 3 | 7 | 12
Not completed — Death | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Progressive Disease | 3 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3 | Total
Number analyzed (Participants) | 24 | 15 | 39 | 78
Age, Continuous [Mean (Full Range); unit: years] | 2 [0 to 12] | 3 [0 to 12] | 7 [0 to 20] | 5 [0 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 27 | 51
  Male | 10 | 5 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 16 | 35
  Not Hispanic or Latino | 9 | 8 | 20 | 37
  Unknown or Not Reported | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 15 | 12 | 28 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 7 | 13
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 2 | 3 | 5
  United States | 12 | 7 | 24 | 43
  Brazil | 12 | 6 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Five Year Event-free Survival (EFS)
Description: The model used for comparison will be an exponential model with a constant failure rate of 0.053 (stratum I), 0.347 (stratum II), 0.602 (stratum III and IV) per year for the first two years and 0 after that. The one-sample one-sided log-rank test comparing the observed data with the hypothesized model (Woolson, 1981) of size 0.05 will be used to assess whether the data are consistent with the target models. Since this test has independent increments, the method of Lan and DeMets will be used to derive the p-values for testing procedure.
Time Frame: Up to five years after enrollment
Measure: Number (95% Confidence Interval); unit: Estimated probability five year EFS
Arm/Group | Stratum 1 | Stratum 2 | Stratum 3
Number analyzed (Participants) | 24 | 15 | 39
Estimated probability five year EFS | 0.86 [0.62 to 0.95] | 0.53 [0.26 to 0.74] | 0.51 [0.33 to 0.66]
Statistical Analysis 1: Comparison: Stratum 1; We will test the 2-year EFS is 90% using the asymptotic distribution of the complementary log-log distribution of the Kaplan-Meier (KM) estimate; Test type: Other; p = 0.44, 2-year KM estimate; 2 Year EFS = 0.89
Statistical Analysis 2: Comparison: Stratum 2; We will test the 2-year EFS is 50% using the asymptotic distribution of the complementary log-log distribution of the Kaplan-Meier (KM) estimate; Test type: Other; p = 0.40, 2-year KM estimate; 2 Year EFS = 0.53
Statistical Analysis 3: Comparison: Stratum 3; We will test the 2-year EFS is 15% using the asymptotic distribution of the complementary log-log distribution of the Kaplan-Meier (KM) estimate; Test type: Other; p = 0.00000853, 2-year KM estimate; 2 Year EFS = 0.55

2. Secondary Outcome: Toxicity Associated With Chemotherapy Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: The proportion of patients assigned to receive chemotherapy that experience CTC Version 4 grade 3 or higher anemia at any time during protocol therapy
Time Frame: Up to 182 Days After Enrollment
Measure: Number; unit: participants
Arm/Group | Stratum 3
Number analyzed (Participants) | 39
participants
  Incidence of Abdominal Infection | 1
  Incidence of Abdominal Pain | 2
  Incidence of Acidosis | 1
  Activated Partial Thromboplastin Time Prolonged | 1
  Incidence of Adrenal Insufficiency | 5
  Incidence of Alanine Aminotransferase Increased | 2
  Incidence of Allergic Reaction | 1
  Incidence of Anemia | 22
  Incidence of Anorexia | 7
  Incidence of Aspartate Aminotransferase Increased | 2
  Incidence of Blood Bilirubin Increased | 1
  Incidence of Cardiac Disorders - Other, Specify | 2
  Incidence of Catheter Related Infection | 3
  Incidence of Colitis | 1
  Incidence of Confusion | 1
  Incidence of Dehydration | 3
  Incidence of Depressed Level of Consciousness | 1
  Incidence of Diarrhea | 1
  Incidence of Dyspnea | 2
  Incidence of Enterocolitis Infectious | 1
  Incidence of Esophagitis | 2
  Incidence of Febrile Neutropenia | 16
  Incidence of Fever | 1
  Incidence of Gastrointestinal Disorders - Other, S | 2
  Incidence of Generalized Muscle Weakness | 1
  Incidence of GGT Increased | 1
  Incidence of Hearing Impaired | 6
  Incidence of Heart Failure | 1
  Incidence of Hyperglycemia | 3
  Incidence of Hyperkalemia | 3
  Incidence of Hypertension | 1
  Incidence of Hypocalcemia | 3
  Incidence of Hypoglycemia | 1
  Incidence of Hypokalemia | 9
  Incidence of Hypomagnesemia | 2
  Incidence of Hyponatremia | 7
  Incidence of Hypophosphatemia | 4
  Incidence of Hypotension | 2
  Incidence of Hypoxia | 3
  Incidence of Infections and Infestations - Other, | 7
  Incidence of INR Increased | 1
  Incidence of Left Ventricular Systolic Dysfunction | 2
  Incidence of Lung Infection | 1
  Incidence of Lymphocyte Count Decreased | 2
  Toxicity Associated with Mitotane | 4
  Incidence of Mucositis Oral | 6
  Incidence of Nausea | 5
  Incidence of Neutrophil Count Decreased | 20
  Incidence of Obstruction Gastric | 1
  Incidence of Pain | 1
  Incidence of Peripheral Motor Neuropathy | 1
  Incidence of Peripheral Sensory Neuropathy | 1
  Incidence of Pharyngitis | 1
  Incidence of Platelet Count Decreased | 20
  Incidence of Pneumonitis | 3
  Incidence of Premature Menopause | 1
  Incidence of Rash Maculo-papular | 1
  Incidence of Sepsis | 2
  Incidence of Skin Infection | 1
  Incidence of Sore Throat | 1
  Incidence of Upper Respiratory Infection | 1
  Incidence of Urinary Tract Infection | 1
  Incidence of Vascular Access Complication | 2
  Incidence of Ventricular Arrhythmia | 1
  Incidence of Vomiting | 5
  Incidence of White Blood Cell Decreased | 16
  Incidence of Wound Infection | 1

3. Secondary Outcome: Complications Associated With Radical Adrenalectomy and RLND
Description: Any patient who dies because of surgery or has a grade 3 or 4 toxicity possibly, probably or likely related to surgery will be considered as having experienced a surgical complication. The complication rate is estimated as the proportion of evaluable patients that have a complication.
Time Frame: Up to 1 month after surgery
Population: Sixty-nine eligible patients received surgery of the primary tumor site or RPLND. Complication rates were considered over the entire population regardless of Arm/Group assignment. One patient had grade 3 abdominal pain attributed to surgery.
Measure: Number; unit: participants
Groups:
- All Patients: The complication rate is estimated as the proportion of evaluable patients that have a complication as it relates to surgery.
Arm/Group | All Patients
Number analyzed (Participants) | 69
participants | 1

4. Secondary Outcome: Frequency of Lymph Node Involvement by Imaging.
Description: The number eligible patients who have lymph node involvement by imaging at study enrollment.
Time Frame: At study enrollment
Population: Seventy-five eligible patients had tumor imaging done at the time of study enrollment and evaluated for the presence of lymph node involvement
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Regardless of Arm/Group assignment, the frequency reflects the total number of patients who had lymph node involvement by imaging at study enrollment.
Arm/Group | All Patients
Number analyzed (Participants) | 75
Participants | 71

5. Secondary Outcome: Incidence and Type of Germline TP53 Mutations in Non-Brazilian Children and Children From Southern Brazil by Deoxyribonucleic Acid (DNA) Sequencing and Affymetrix Gene Chip Analysis.
Description: The proportion of patients in each subpopulation are compared.This test is dependent on the number of patients from whom blood can be obtained as well as the frequency of the relevant mutation in each group.
Time Frame: At study enrollment
Population: The proportion of patients in each subpopulation are compared.This test is dependent on the number of patients from whom blood can be obtained as well as the frequency of the relevant mutation in each group (Number of patients from Brazil: 23. Number of patients not from Brazil: 31)
Measure: Number; unit: participants
Groups:
- All Patients: Regardless of Arm/Group assignment, the number of eligible patients from whom blood was obtained as well as the frequency of the relevant mutation in each group.
Arm/Group | All Patients
Number analyzed (Participants) | 54
participants
  C229R mutation in p53 in Patients from Brazil | 0
  C229R mutation in Patients not from Brazil | 2
  E180K mutation in p53 in Patients from Brazil | 0
  E180K mutation in Patients not from Brazil | 1
  G245C mutation in p53 in Patients from Brazil | 0
  G245C mutation in Patients not from Brazil | 1
  I254T mutation in p53 in Patients from Brazil | 1
  I254T mutation in Patients not from Brazil | 0
  L265Q mutation in p53 in Patients from Brazil | 0
  L265Q mutation in Patients not from Brazil | 1
  P47S mutation in p53 in Patients from Brazil | 0
  P47S mutation in Patients not from Brazil | 1
  Q52fs mutation in p53 in Patients from Brazil | 0
  Q52fs mutation in Patients not from Brazil | 1
  R158L mutation in Patients from Brazil | 0
  R158L mutation in Patients not from Brazil | 1
  G245S mutation in Patients from Brazil | 0
  G245S mutation in Patients not from Brazil | 1
  R213P mutation in p53 in Patients from Brazil | 0
  R213P mutation in Patients not from Brazil | 1
  R248L mutation in Patients from Brazil | 0
  R248L mutation in Patients not from Brazil | 1
  R282W mutation in p53 in Patients from Brazil | 0
  R282W mutation in p53 in Patients not from Brazil | 1
  R283H mutation in p53 in Patients from Brazil | 0
  R283H mutation in p53 in Patients not from Brazil | 31
  R337H mutation in p53 in Patients from Brazil | 20
  R337H mutation in p53 in Patients not from Brazil | 0
  R342X mutation in p53 in Patients from Brazil | 0
  R342X mutation in p53 in Patients not from Brazil | 1
  T125T c375G>A muation in p53 in Pts from Brazil | 1
  T125T c375G>A mutation in p53 in pts not from Braz | 1
  T125T splice in DBD in pts from Brazil | 0
  T125T splice in DBD in pts not from Brazil | 1
  wild type p53 in Patients from Brazil | 1
  wild type p53 in Patients not from Brazil | 16

6. Secondary Outcome: Molecular Alterations and Embryonal Markers in Children With ACT - A43 del33bp Mutation of (Beta)-Catenin.
Description: The number of eligible patients who have A43 del33bp mutation of (beta)-catenin.
Time Frame: Patients who had surgery at time of enrollment.
Population: Fifty-eight eligible patients had material examined for the presence of (beta)-catenin mutations.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: Regardless of Arm/Group assignment, the number of eligible patients who had surgery at study enrollment and have A43 del33bp mutation of (beta)-catenins.
Arm/Group | All Patients
Number analyzed (Participants) | 58
Participants
  children with ACT - wild type (beta)-catenin | 51
  A43 del33bp mutation of (beta)-catenin | 1

7. Secondary Outcome: Frequency of Tumor Spillage at the Time of Tumor Resection
Description: The number of eligible patients who have surgical resection of the primary tumor and have tumor spillage at the time of resection.
Time Frame: Up to one year or while on protocol therapy, whichever is less
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: The number of eligible patients who have surgical resection of the primary tumor and have tumor spillage at the time of resection.
Arm/Group | All Patients
Number analyzed (Participants) | 69
Participants | 15

ADVERSE EVENTS:
Description: Serious and other adverse events were collected only for Stratum 3 patients who received systemic intervention. Stratum 1 and Stratum 2 patients did not receive chemotherapy as part of protocol treatment.
Arm/Group | Stratum 3
Serious Adverse Events (participants affected / at risk) | 1/39
Other Adverse Events (participants affected / at risk) | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 3 (N=39)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 3 (N=39)
Abdominal infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 5 (5)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 24 (24)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3)
Catheter related infection (Infections and infestations) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (16)
Fever (General disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
GGT increased (Investigations) | 1 (1)
Growth suppression (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 9 (9)
Heart failure (Cardiac disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypertension (Vascular disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 9 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 7 (7)
INR increased (Investigations) | 1 (1)
Irritability (General disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3)
Malaise (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (6)
Neutrophil count decreased (Investigations) | 20 (20)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 21 (21)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Precocious puberty (Endocrine disorders) | 1 (1)
Premature menopause (Reproductive system and breast disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Retinal vascular disorder (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 16 (16)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.